CLINICAL TRIAL: NCT05389605
Title: A Single Centre Experience of Local Perforator Flaps in Oncoplastic Breast Surgery; a Cross-sectional Study
Brief Title: Outcomes of Local Perforator Flaps in Oncoplastic Surgery
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Sana Zeeshan, Assistant Professor, Aga Khan University
Other Study IDs: ERC#2020-3379-10190
Record Dates: First submitted 2022-05-10; First posted 2022-05-25 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Breast Tumor; Perforator Flap; Breast Cancer; Oncoplasty; Breast-Q
Keywords: Local Perforator Flaps; Breast Cancer; Oncoplastic Breast Conserving Surgery; BREAST-Q; Breast Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention was undertaken — This was an observational study, no intervention was done.

SUMMARY:
This is a single center experience of using local perforator flaps in partial breast reconstruction for breast tumors while evaluating cosmetic outcomes, patient satisfaction and well-being using a validated self-administered questionnaire.

DETAILED DESCRIPTION:
Background & Objectives: Various oncoplastic techniques have emerged over the years to preserve breast cosmesis and symmetry without compromising the principles of tumor excision. One of the newer techniques for breast volume replacement to achieve symmetry and cosmesis is the use of fasciocutaneous pedicled chest wall perforator flaps or local perforator flaps (LPF). The objectives of this study are to document the details of the surgical procedure as well as patient-reported satisfaction and well-being following the already performed surgical procedure using a validated BREAST-Q tool among Pakistani women.

Materials & Methods: This prospective cross-sectional study will be conducted by enrolling all the 25 female patients who have undergone LPF for breast tumors at The Aga Khan University Hospital, Karachi. Data related to the procedure will be collected on a pre-designed proforma. Cosmetic outcomes and patient satisfaction will be evaluated using 2 scales from BREAST-Q BCT domain version 2.0. The questionnaire will be self-administered by the patients during their routine follow-up in the clinic. Data will be analyzed using the Statistical Package for Social Sciences (SPSS) version 23. Mean (SD) / median (IQR) will be computed for quantitative variables and frequency and percentages will be calculated for qualitative variables. 2 sample t-test will be applied. P-value ≤0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All female patients suitable for breast conservation who underwent a pedicled fasciocutaneous perforator flap for immediate partial breast reconstruction at the breast surgery section

Exclusion Criteria:

* For evaluation of surgical techniques, since this was a review of cases already operated, no cases were excluded.
* For cosmetic outcomes and patient satisfaction, patients who lost to follow, expired or did not give consent to participate in the study were excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All female patients who underwent a pedicled fasciocutaneous perforator flap for immediate partial breast reconstruction in the Breast section of The Aga Khan University Hospital were included in the study. For cosmetic outcomes and patient satisfaction, a follow-up of at least 3 months after surgery before participation in the survey was mandatory.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical techniques of pedicled local fasciocutaneous perforator flaps in partial breast reconstruction in terms of flap anatomy | May 2018 to February 2021
  Flap anatomy involves the type of flap
Surgical techniques of pedicled local fasciocutaneous perforator flaps in partial breast reconstruction in terms of location of perforators | May 2018 to February 2021
Surgical techniques of pedicled local fasciocutaneous perforator flaps in partial breast reconstruction in terms of operative time | May 2018 to February 2021
Surgical techniques of pedicled local fasciocutaneous perforator flaps in partial breast reconstruction in terms of post-operative morbidities | May 2018 to February 2021

SECONDARY OUTCOMES:
Cosmetic outcomes of patients following local perforator flaps in oncoplastic breast conserving surgery | April 2020 to June 2021
  Cosmetic outcomes will be measured using the validated BREAST-Q Breast-Conserving Therapy (BCT) domain version 2.0. Patient's answers are converted to a number from 0 (worst) to 100 (best) using the Q-Score tool.
Patient satisfaction following local perforator flaps in oncoplastic breast conserving surgery | April 2020 to June 2021
  Patient satisfaction will be measured using the validated BREAST-Q Breast-Conserving Therapy (BCT) domain version 2.0. Patient's answers are converted to a number from 0 (worst) to 100 (best) using the Q-Score tool.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Zeeshan, FCPS, FACS, Principal Investigator — Aga Khan University
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher B, Anderson S, Redmond CK, Wolmark N, Wickerham DL, Cronin WM. Reanalysis and results after 12 years of follow-up in a randomized clinical trial comparing total mastectomy with lumpectomy with or without irradiation in the treatment of breast cancer. N Engl J Med. 1995 Nov 30;333(22):1456-61. doi: 10.1056/NEJM199511303332203. PMID 7477145
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Esser JFS. Biological- or artery flaps of the face [Internet]. Monaco: Institut Esser de Chirurgie Structive; 1931 [cited 2022 Apr 27]. Available from: https://wellcomecollection.org/works/pf3qfx2r/items?canvas=7
- [Background] Hamdi M, Van Landuyt K, de Frene B, Roche N, Blondeel P, Monstrey S. The versatility of the inter-costal artery perforator (ICAP) flaps. J Plast Reconstr Aesthet Surg. 2006;59(6):644-52. doi: 10.1016/j.bjps.2006.01.006. Epub 2006 Mar 22. PMID 16716957
- [Background] Hamdi M, Van Landuyt K, Monstrey S, Blondeel P. Pedicled perforator flaps in breast reconstruction: a new concept. Br J Plast Surg. 2004 Sep;57(6):531-9. doi: 10.1016/j.bjps.2004.04.015. PMID 15308400
- [Background] Losken A, Hamdi M. Partial breast reconstruction: current perspectives. Plast Reconstr Surg. 2009 Sep;124(3):722-736. doi: 10.1097/PRS.0b013e3181b179d2. PMID 19730292
- [Background] McCulley SJ, Schaverien MV, Tan VK, Macmillan RD. Lateral thoracic artery perforator (LTAP) flap in partial breast reconstruction. J Plast Reconstr Aesthet Surg. 2015 May;68(5):686-91. doi: 10.1016/j.bjps.2015.01.008. Epub 2015 Jan 27. PMID 25660559
- [Background] BREAST-Q ® VERSION 2.0 © Memorial Sloan Kettering Cancer Center and The University of British Columbia, 2017. All rights reserved
- [Background] Pusic A, Klassen A, Cano S. BREAST-Q Version 2.0 © A Guide for Researchers and Clinicians [Internet]. 2017 [cited 2022 Apr 27]. Available from: https://qportfolio.org/wp-content/uploads/2018/12/BREAST-Q-USERS-GUIDE.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT05389605/Prot_SAP_000.pdf